CLINICAL TRIAL: NCT05321797
Title: Effects Of Aerobic Training On Spasticity And Gross Motor Function In Children With Diplegic Cerebral Palsy
Brief Title: Aerobic Training On Spasticity And Gross Motor Function In Children With Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/0702
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Palsy
Keywords: Aerobic Training; Gross Motor Function; Stationary Cycle; Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training Group (Experimental): Cycling exercise group along with Conventional therapy
  Interventions: Other: Aerobic Training; Other: Conventional Physiotherapy
- Conventional Physiotherapy (Active Comparator): Strectching with ROM and gait training
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Aerobic Training — This group will be administered with the cycling exercises in addition to the complete plan of care that is being administered to the control group. The cycling intervention will be performed 3 times per week, for 30 minutes, within a 12-week period
  Arms: Aerobic Training Group
Other: Conventional Physiotherapy — This group will be administered with Conventional Physiotherapy that includes 5 minutes of stretching exercises for quadriceps, hamstrings and gastrocnemius, 5 minutes of trunk control training, 5 minutes walking in the hall with and without the therapist assistance, walker or crutches, and finally 5 minutes of breathing exercises for Relaxation

SUMMARY:
To determine the effects of aerobic training on spasticity and gross motor function in children with diplegic Cerebral palsy.Cerebral palsy (CP) is a neurodevelopmental disorder characterized by abnormalities of muscle tone, movement and motor skills, and is attributed to injury to the developing brain. . The spastic CP is found to be the commonest presentation followed by athetoid, ataxic and mixed types. Children with cerebral palsy (CP) have decreased capacity to participate in play and sports activities .Reduced capacity to perform typical childhood activities contributes to low habitual physical activity and declining gross motor function in adolescence. Exercise opportunities are restricted in the population of cerebral palsy with spasticity, and so muscle strength may be reduced by disuse. Aerobic Training via Lower-extremity cycling is a rehabilitation tool used by physical therapists to improve spasticity, gross motor function and cardio-respiratory fitness, appears well-suited as a therapeutic intervention for children with CP. The tools used will be GMFM-66 and Modified Ashworth Scale. Study will be conducted on Thirty two patients in two Groups. Group A will be Control Group that will be provided with conventional physiotherapy (Stretching exercises , Trunk control training, walk and breathing exercises) and Group B will be Experimental Group that will be provided with conventional physiotherapy with cycling for 30 minutes with three sessions per week over the period of 12 weeks. Data will be analyzed using spss 22.0.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years of age both genders will be included.
* Ability to follow simple verbal instructions.
* Ability to walk independently, with or without an assistive device, for short distances (gross motor function classification system [gmfcs] levels i-iii)
* Spastic Diplegic Cerebral Palsy scoring on Ashworth Scale of 1, 1±, 2

Exclusion Criteria:

* Orthopedic surgery, neurological surgery, or baclofen pump implantation within the preceding 12 months
* Botulinum toxin injections within the preceding 3 months
* Serial casting or new orthotic devices within the preceding 3 months
* Initiation of oral medications that affect the neuromuscular system (eg, baclofen) within the preceding 3 months
* Inability or unwillingness to maintain age appropriate behavior
* Serious medical conditions such as cardiac disease, diabetes, or uncontrolled seizures
* Significant hip, knee, or ankle joint contractures preventing passive movement of the lower limbs through the pedaling cycle

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-66) | 8th Week
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline. However, most of the items have specific descriptors for each score. It is imperative that the guidelines contained in the manual be used for scoring each item. SCORING KEY 0 = does not initiate 1 = initiates 2 = partially completes 3 = completes 9 (or leave blank) = not tested (NT).
Modified Ashworth Scale (MAS) | 8th week
  The modified Ashworth scale(MAS) is a 6-point rating scale that is used to measure muscle tone.(20) The reliability of the modified Ashworth scale was very good reliability and validity

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Physiogic Physiotherapy Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damiano DL, Stanley CJ, Ohlrich L, Alter KE. Task-Specific and Functional Effects of Speed-Focused Elliptical or Motor-Assisted Cycle Training in Children With Bilateral Cerebral Palsy: Randomized Clinical Trial. Neurorehabil Neural Repair. 2017 Aug;31(8):736-745. doi: 10.1177/1545968317718631. Epub 2017 Jul 8. PMID 28691601
- [Background] Fowler EG, Knutson LM, Demuth SK, Siebert KL, Simms VD, Sugi MH, Souza RB, Karim R, Azen SP; Physical Therapy Clinical Research Network (PTClinResNet). Pediatric endurance and limb strengthening (PEDALS) for children with cerebral palsy using stationary cycling: a randomized controlled trial. Phys Ther. 2010 Mar;90(3):367-81. doi: 10.2522/ptj.20080364. Epub 2010 Jan 21. PMID 20093327
- [Background] Fujimoto J, Umemoto Y, Koike Y, Isida K, Sakamoto K, Tajima F. Immediate effects of short period lower limb ergometer exercise in adolescent and young adult patients with cerebral palsy and spastic diplegia. J Phys Ther Sci. 2021 Jan;33(1):52-56. doi: 10.1589/jpts.33.52. Epub 2021 Jan 5. PMID 33519075
- [Background] da Rosa Pinheiro DR, Cabeleira MEP, da Campo LA, Correa PS, Blauth AHEG, Cechetti F. Effects of aerobic cycling training on mobility and functionality of acute stroke subjects: A randomized clinical trial. NeuroRehabilitation. 2021;48(1):39-47. doi: 10.3233/NRE-201585. PMID 33386826
- [Background] El-Tamawy MS, Darwish MH, Basheer MA, Reda AM, Elzanaty M, Khalifa HA. Effect of cycling exercise on motor excitability and gait abnormalities in stroke patients. The Egyptian Journal of Neurology, Psychiatry and Neurosurgery. 2021;57(1):1-7
- [Background] Armstrong EL, Spencer S, Kentish MJ, Horan SA, Carty CP, Boyd RN. Efficacy of cycling interventions to improve function in children and adolescents with cerebral palsy: a systematic review and meta-analysis. Clin Rehabil. 2019 Jul;33(7):1113-1129. doi: 10.1177/0269215519837582. Epub 2019 Apr 2. PMID 30935240